CLINICAL TRIAL: NCT03162887
Title: Mammogram Decision Support for Formerly Homeless Women With Serious Mental Illness
Brief Title: Educational Module and Decision Counseling Program in Increasing Mammography Screening Rates in Formerly Homeless Women With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14G.62; JT 6000 (Other: JeffTrial Number); 123369-CCCDA-12-213-01-CC (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast - Female
MeSH Terms: interventions — Early Intervention, Educational; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (education module, counseling) (Experimental): Participants receive a research team member-led breast cancer and mammogram educational module and undergo a web-based decision counseling session over 2 hours. Participants then receive a "next steps" document and may undergo an interview to discuss their decision-making process and relevant experiences during the course of the study.
  Interventions: Other: Educational Intervention; Other: Counseling; Other: Informational Intervention

INTERVENTIONS:
Other: Educational Intervention — Receive a research team member-led breast cancer and mammogram educational module
  Other Names: Intervention through Education
Other: Counseling — Undergo a web-based decision counseling session
  Other Names: Counseling Intervention
Other: Informational Intervention — Receive a "next steps" document

SUMMARY:
This pilot clinical trial studies how well an educational module and decision counseling program works in increasing mammography screening rates in formerly homeless women with serious mental illness. An educational module and decision counseling program may be an effective tool and have the potential to help with early detection and treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Increase mammography screening rates in women age 40 and over with experiences of homelessness and serious mental illness (SMI).

II. Increase knowledge, decease psychological distress, and advance decision stage and intention to get a mammogram in study participants.

ELIGIBILITY:
Inclusion Criteria:

* 30 formerly homeless women with a diagnosis of a serious mental illness in the Pathways to Housing or Project HOME supportive housing programs
* Only women that have never received a mammogram are eligible to participate (self-report)
* Participants must be willing to participate in all aspects of research

Exclusion Criteria:

* Participants cannot be decisionally impaired, actively psychotic, or have unstable mental illness that prevents participation in the decisional counseling session
* Women who have had a mammogram will be excluded from the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2014-07-12 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Change in decisional conflict score assessed by pre- and post-intervention survey | Baseline up to 1 month
  Will estimate the mean pre/post change, along with a 95% confidence interval, and will test this change via a paired t-test. Will use linear regression to assess what factors (including socio-demographics and decision counseling score) are associated with the change.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Weinstein, MD, MPH, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/